CLINICAL TRIAL: NCT02535299
Title: The Correlation Between Par-4 and Telomere-telomerase System in the New Dignosised Type 2 Diabetes Patients Who Received GLP-1 Analog or Metformin Treatment
Brief Title: Par-4 and Telomere-telomerase System in Type 2 Diabetes Patients Who Received GLP-1 or Metformin Treatment
Acronym: Par-4；GLP-1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Wu Qinan, the Third Military Medical University, Third Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLP-1
Record Dates: First submitted 2015-08-21; First posted 2015-08-28 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: GLP-1；Metformin；Telomere-telomerase System；Par-4
Keywords: telomere-telomerase; Par-4; GLP-1; metformin
MeSH Terms: interventions — Liraglutide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- insulin (Experimental): basic insulin treatment：glargine 10-30 units once a day based on the glucose control for 6 months.
  Interventions: Drug: Liraglutide; Drug: Metformin

INTERVENTIONS:
Drug: Liraglutide — GLP-1 analog (1.2mg-1.8mg/day) treatment for 6 months
  Other Names: Victoza
Drug: Metformin — Metformin(1500mg-2000mg/day) treatment for 6 months
  Other Names: Glucophage

SUMMARY:
Objectives: To investigate the treatment effect between insulin,metformin and Liraglutide; in Type 2 Diabetes in our hospital, in order to investigate the possible mechanism about telomere-telomerase system and Par-4.

DETAILED DESCRIPTION:
160 Type 2 diabetes in our hospital will divide into 4 groups: group A (40 healthy volunteers), group B (40 patients who give basal and insulin treatment, group C（40 patients who give basal and Liraglutide treatment),group D（40 patients who give basal and metformin treatment). The age, height, weight, blood glucose, glycosylated hemoglobin A1c（HbA1c）,homeostasis model assessment(HOMA-IR), lipid, blood pressure, course of disease, telomere length,telomerase activity will record respectively. And High-sensitive C-reactive protein (HsCRP), Par-4, GST,SOD,GSH-PX,ATF-6,CHOP,XBP-1 and Tumor necrosis factor-α（TNF-α） will detect as Baseline. After each group's treatment, Change from baseline of all indexes will record, Multifactor logistic regression will be analyzed the correlations between each positive indexes.

ELIGIBILITY:
Inclusion Criteria:

* Newly dignosised type 2 diabetes according to WHO criteria.glycated hemoglobin (HbA1c) was more than 10%;
* Seronegative for antibodies against insulin, islet cells and glutamic acid decarboxylase (GAD);

Exclusion Criteria:

* Type 1 diabetes mellitus,presence of autoimmune diabetes indicated by antibodies to insulin, islet cells, and GAD；
* Gestational diabetes;
* patients with heart, liver, or renal function impairment;presence of severe infections or cerebrovascular disease;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
physiological parameter:glycosylated hemoglobin A1c | up to 6 months;
  up to 6 months;;HbA1c was measured by a certified hospital laboratory according to established and approved protocols

SECONDARY OUTCOMES:
physiological parameter:the concentration of Par-4 | up to 6 months;
  up to 6 months;;secretary Par-4 were detected with Par-4 ELISA kit (MBL, USA)
physiological parameter:telomere length | up to 6 months;
  up to 6 months;;Telomere length was measured via fluorescence in situ hybridization using flow cytometry
physiological parameter:telomease activity | up to 6 months;
  up to 6 months;;Telomerase activity was measured using the TeloTAGGG Telomerase PCR ELISAPLUS kit (Roche Diagnostics, Mannheim, Germany)
physiological parameter:TNF-α | up to 6 months;
  up to 6 months, TNF-a levels were measured by commercial ELISA kit following the manufacturer's instructions;TNF-a levels were measured by commercial ELISA kit following the manufacturer's instructions;(MBL, USA)

CONTACTS AND LOCATIONS:
Locations (1):
- Southwest Hospital of the Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided